CLINICAL TRIAL: NCT02242253
Title: A Randomised, Double-blind, Double-dummy, Crossover Efficacy and Safety Comparison of 6-week Treatment Periods of the Free Combinations of Tiotropium Inhalation Powder Capsule (18 μg) QD + Salmeterol Metered Dose Inhaler (2 Puffs of 25 μg) QD or BID, Tiotropium Inhalation Powder Capsule (18 μg) QD and Salmeterol Metered Dose Inhaler (2 Puffs of 25 μg) BID in Patients With (COPD)
Brief Title: Free Combinations of Tiotropium Inhalation Powder Capsule + Salmeterol Metered Dose Inhaler, Tiotropium Inhalation Powder Capsule and Salmeterol Metered Dose Inhaler in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.7
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (4):
- Tiotropium+salmeterol QD (Experimental): free combination of tiotropium and salmeterol
  Interventions: Drug: Tiotropium; Drug: Salmeterol; Drug: Placebo-MDI
- Tiotropium+salmeterol BID (Active Comparator): free combination of tiotropium and salmeterol
  Interventions: Drug: Tiotropium; Drug: Salmeterol; Drug: Placebo-MDI
- Tiotropium QD (Active Comparator)
  Interventions: Drug: Tiotropium; Drug: Placebo-MDI
- Salmeterol BID (Active Comparator)
  Interventions: Drug: Salmeterol; Drug: Placebo HandiHaler®

INTERVENTIONS:
Drug: Tiotropium — administered via HandiHaler®
  Arms: Tiotropium QD; Tiotropium+salmeterol BID; Tiotropium+salmeterol QD
Drug: Salmeterol — administered via metered dose inhaler (MDI)
  Arms: Salmeterol BID; Tiotropium+salmeterol BID; Tiotropium+salmeterol QD
Drug: Placebo-MDI
  Arms: Tiotropium QD; Tiotropium+salmeterol BID; Tiotropium+salmeterol QD
Drug: Placebo HandiHaler®
  Arms: Salmeterol BID

SUMMARY:
Main Study: To evaluate and to compare the lung function response to the free combinations of tiotropium 18 μg (QD) + salmeterol 50 μg (QD or BID), salmeterol 50 μg BID and tiotropium 18 μg QD at the end of 6-week treatment periods in patients with COPD.

Sub-Study: Was performed in subset of patients participating in the Main Study to assess the effect of the four randomised treatments on dynamic hyperinflation.

Extension Study: To establish whether the FEV1 time profile following combination bronchodilator therapy of tiotropium plus salmeterol is affected by the pharmaceutical formulation of salmeterol, i.e. the MDI or the Diskus®.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 ≤ 60% of predicted normal and FEV1 ≤ 70% of FVC (Visits 1 and 2)
3. Male or female patients 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years (Patients who had never smoked cigarettes have to be excluded)
5. Patients must be able to perform technically acceptable pulmonary function tests and must be able to maintain records (Patient Daily Diary Card) during the study period as required in the protocol
6. Patients must be able to inhale medication in a competent manner from the HandiHaler® device and from a metered dose inhaler (MDI)

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis, if the abnormality defines a significant disease as defined in exclusion criterion No. 1
3. Patients with a recent history (i.e. six months or less) of myocardial infarction
4. Patients with any unstable or life-threatening cardiac arrhythmia or patients who have been hospitalised for such an event within the past year
5. Patients with a malignancy for which the patient has undergone resection, Radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed
6. Patients with known narrow-angle glaucoma
7. Patients with a history of asthma, allergic rhinitis or who have a total blood eosinophil count ≥600 mm3
8. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
9. Patients with known active tuberculosis
10. Patients with a history of and/or active significant alcohol or drug abuse. See exclusion criterion No. 1
11. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1
12. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1)
13. Patients who regularly use daytime oxygen therapy
14. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
15. Patients who are being treated with oral beta-adrenergics
16. Patients who are being treated with cromolyn sodium or nedocromil sodium
17. Patients who are being treated with antihistamines (H1 receptor antagonists), antileukotrienes or leukotriene receptor antagonists for asthma or excluded allergic conditions. See exclusion criterion No. 7
18. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
19. Patients with known hypersensitivity to anticholinergic drugs, beta-adrenergics, lactose or any other components of the medication delivery systems
20. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous 3 months (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants eg: Norplant®)
21. Patients with previous participation (receipt of randomised treatment) in this study
22. Patients who are currently participating in another study
23. The randomisation of patients with any respiratory infection or COPD exacerbation in the six weeks prior to the Screening Visit (Visit 1) or during the baseline period should be postponed. Patients may be randomised six weeks following recovery from the infection or exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2003-09; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve of forced expiratory volume in one second (FEV1 AUC0-24h) | up to 12 hours after morning and evening dose
FEV1 AUC0-12h | up to 12 hours after morning and evening dose

SECONDARY OUTCOMES:
FEV1 AUC12-24h | after 6 weeks of each treatment
AUC of forced vital capacity (FVC AUC0-12h) | after 6 weeks of each treatment
FVC AUC0-24h | after 6 weeks of each treatment
FVC AUC12-24h | after 6 weeks of each treatment
Peak FEV1 | after 6 weeks of each treatment
Trough FEV1 | after 6 weeks of each treatment
  Trough FEV1 was defined as the pre-dose FEV1 measured just prior to the last administration of the morning dose of randomised treatment.
Peak FVC | after 6 weeks of each treatment
Trough FVC | after 6 weeks of each treatment
  Trough FVC was defined as the pre-dose FVC measured just prior to the last administration of the morning dose of randomised treatment
Individual FEV measurements at each time point | up to 6 weeks
Individual FVC measurements at each time point | up to 6 weeks
Peak expiratory flow rate (PEFR) measured twice daily | weeks 4 to 6 of each treatment period
Number of inhalations of rescue salbutamol therapy used per day | weeks 4 to 6 of each treatment period
Change in focal score of the Mahler Transition Dyspnea Index (TDI) | after 6 weeks of each treatment
  The TDI focal score is the sum of the three components of the TDI: Functional Impairment, Magnitude of Task and Magnitude of Effort
Number of patients with adverse events | up to 33 weeks